CLINICAL TRIAL: NCT05206812
Title: Window of Opportunity Trial of Durvalumab (MEDI4736) to Identify Immune Dynamics in Operable Non-small Cell Lung Cancer (NSCLC) (MIRACLE)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1621
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- durvalumab (Experimental): The operable non-small cell lung carcinoma patients (resectable stage IIA~IIIB)
  Interventions: Drug: durvalumab

INTERVENTIONS:
Drug: durvalumab — * durvalumab 1500 mg QD*
  * Surgery within 1 to 8 weeks - 4 cycles of durvalumab 1500 mg/m2 (Day 1, Day 8)+cisplatin 80 mg/m2 (Day 1) q3wks -durvalumab 1500 mg q4wks (Maximum of 10 cycles)

SUMMARY:
This study is phase II, open label, clinical trial of durvalumab to identify immune dynamics in operable non-small cell lung cancer.

DETAILED DESCRIPTION:
In this study, the investigators plan to administer neoadjuvant durvalumab and adjuvant durvalumab to the operable NSCLC patients (resectable stage IIA~IIIB) regardless of PD-L1 status.

Durvalumab 1500mg IV will be administered once prior to surgery. Within 1-8 weeks after completion of durvalumab, patients will undergo surgery. Regardless of MRD status, patients will receive adjuvant treatment of durvalumab 1500mg IV q3 weeks with SoC platinum-based chemotherapy for a total of 4 cycles.

** Adjuvant chemotherapy will be based on standard of care treatment: navelbine 20mg/m2 (D1, 8) and cisplatin 80mg/m2 (D1) (q3w x 4 cycles).

Thereafter, patients will be administered with adjuvant durvalumab 1500mg IV q4 weeks for 10 cycles

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed operable NSCLC (resectable stage IIA~IIIB) regardless of PD-L1 expression.
2. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to neoadjuvant durvalumab.
3. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Male or female, 18 years or older (at the consent is obtained). Note: In the Republic of Korea, a participant must be over 19 years of age inclusive, at the time of signing the informed consent.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Life expectancy of > 12 weeks
7. Body weight >30 kg
8. Adequate normal organ and marrow function as defined below:

   Hemoglobin ≥9.0 g/dL Absolute neutrophil count (ANC) ≥1.0 × 109 /L Platelet count ≥75 × 109/L Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.

   AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN

   Measured creatinine clearance (CL) >60 mL/min or Calculated creatinine CL>60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) / 72 x serum creatinine (mg/dL) x 0.85
9. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
10. Must have a life expectancy of at least 12 weeks

Exclusion Criteria:

1. Patients with EGFR mutations (identified with local testing).
2. Any prior treatment for NSCLC, including prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody, chemo, RT, target therapy or investigational drug.
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
4. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria A. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

   B. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
5. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
6. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
7. History of allogenic organ transplantation.
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   A. Patients with vitiligo or alopecia B. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement C. Any chronic skin condition that does not require systemic therapy D. Patients without active disease in the last 5 years may be included but only after consultation with the study physician E. Patients with celiac disease controlled by diet alone
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
10. History of another primary malignancy except for A. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence B. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease C. Adequately treated carcinoma in situ without evidence of disease
11. History of leptomeningeal carcinomatosis
12. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart). Patient safety and the cardiac SKG should be consulted as needed.
13. History of active primary immunodeficiency
14. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis CPatients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
15. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    A. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) B. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent C. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
16. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
17. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
19. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
20. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | Right after the surgery
  Evaluate the pathologic response in resected tumor tissue. The major pathologic response is defined as less than 10% viable tumors after treatment.

SECONDARY OUTCOMES:
Minimal residual disease | At screening, Post neo-adjuvant durvalamab (+ 1 week ~ prior to surgery), Post-op (3-4 weeks after surgery), Post-op at 3 months (+/- 7 days), Post-op at 6 months (+/- 7 days), After progression (+/- 7 days)
Locoregional control | UP to 2years
Distant metastases free survival | UP to 3years
Disease-free survival | UP to 3years
Overall survival (OS) | Up to 5years

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Hye Ryun, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No